CLINICAL TRIAL: NCT02627482
Title: The Feasibility of Employing Ambulatory Fetal Heart Rate Monitoring in Small for Gestational Age Fetuses at Risk of Stillbirth.
Brief Title: Ambulatory Fetal Heart Rate Monitoring in Small Babies
Status: Completed | Type: Observational
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Habiba Kapaya, Clinical Lecturer, Sheffield Teaching Hospitals NHS Foundation Trust
Other Study IDs: STH18636
Record Dates: First submitted 2015-11-21; First posted 2015-12-11 (Estimated); Last update posted 2017-05-01 (Actual); Status verified 2017-04

CONDITIONS: High Risk Pregnancy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Fetal heart rate monitor (Monica AN24) — The AN24 is a portable, battery powered device, developed in the UK and designed to monitor passively an unborn baby in the antenatal period. The device is CE marked and is attached via a cable assembly which in turn attaches to five standard disposable electrodes placed on the abdomen of a pregnant woman. It is intended for ambulatory use in either the home or hospital environment.
  The AN24 has had rigorous checks in the UK and has been used in many European countries. No hazards have been identified that could compromise the safety of, or cause harm to the fetus or the mother. The only potential issue identified is a local reaction under the electrodes. Nonetheless, the electrodes used are the standard disposable ECG electrodes, used routinely for adult ECG measurements.

SUMMARY:
Most babies who measure small during pregnancy are born healthy. However, some are small because they are not growing as expected, usually because the placenta (the baby's 'life support' system) is not working properly. These babies are at greatly increased risk of dying before birth, and need to be delivered before they become poorly.

Scans and electronic heartrate monitoring are currently used to monitor these babies. But they can only be used for short periods and don't always provide enough information to show when to deliver the baby.

A small light monitor has been developed that safely records the baby's heart rate for up to 16hrs by measuring electrical activity through sticky patches on the mum's skin (like a normal ECG). The woman carries on with her daily activities while wearing it. Monitoring the heart rate over a longer time may help with decisions about the timing of the delivery and could prevent stillbirth, the aim of our future study. This will include large numbers of women carrying small babies. Before the investigators can do this the investigators need to know whether:

1. Wearing the monitor for 16hrs is practical and acceptable to pregnant women
2. The monitor can provide useful information on the baby's heart rate at different stages of pregnancy.

Thirty pregnant women whose babies are measuring small will be asked to wear the monitor on two occasions, for 16hrs each time. The women will describe what they think about wearing the monitor by completing questionnaires.

The data from the monitor will be downloaded and compared with the woman's medical notes after the participant has delivered her baby. Results from this study will be publicised and will help with the design of the investigators future study into the usefulness of this monitor.

DETAILED DESCRIPTION:
Study design:

The study has been designed as a prospective, non randomised, single centre feasibility study to determine the acceptability and reliability of the Monica AN24 device, as a method of long-term fetal heart rate (FHR) monitoring on more than one occasion in the antenatal period.

Objectives of the study:

The proposed feasibility study aims to:

1. Assess the recruitment rates and practicality of the study design and protocol.
2. Evaluate the acceptability to participants of wearing the device for overnight FHR monitoring on two occasions in pregnancy.
3. Measure the success rate of generating good quality overnight FHR data and identify any limitations of the technique.
4. Determine response rates to questionnaires

Recruitment The investigators will recruit women from 28 completed weeks of gestation. The investigators will study each participant on two occasions (2-4 weeks apart). Being a feasibility study FHR data obtained during these experiments will not be employed in the routine clinical care of study participants whose care will follow standard patterns of surveillance employed at the Jessop Wing Hospital (JW), Sheffield.

Statistical analysis:

As this is a feasibility study the investigators will employ mainly descriptive analysis. The investigators will report rates of consent, recruitment and acceptability of wearing the AN24 device on two occasions. The investigators shall also report the rates and duration of obtaining valid FHR data when the device is worn. The feasibility and FHR outcome measures will be summarised and will inform design for future definitive studies.

Future work and clinical impact of this research:

The investigators believe that incorporating ambulatory FHR monitoring to the current methods employed to monitor SGA could predict and prevent stillbirth. This is the overarching aim of our future definitive multicentre study which will require collection of longterm FHR data at different stages of pregnancy from at least 500 women carrying small babies. Data captured from our feasibility study will inform the design of our main study and ensure that our design is robust and that all the potential issues identified in the feasibility study have been addressed.

ELIGIBILITY:
Inclusion Criteria:

All women with singleton pregnancy from 28 completed weeks of gestation, suspected to carry small for gestational age (SGA) fetus on ultrasound scan but with no known congenital abnormality will be eligible for inclusion in the study if they agree.

Exclusion Criteria:

* Evidence of a major fetal malformation on ultrasound scan
* Clinical suspicion of labour
* Multiple pregnancy
* Involved in another study using a device or medicinal product

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The Investigators will recruit 30 women with a singleton pregnancy (no congenital abnormality) and a customised birth weight ratio of less than 10th centile on ultrasound from the small baby clinic, which is provided at the Fetomaternal Unit (FMU) at the Jessop Wing (JW) Hospital, Sheffield. Each participant will be studied on 2 occasions, 2 to 4weeks apart at their routine hospital visit for serial ultrasound scans.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2015-09; Primary Completion 2016-11-08 (Actual); Study Completion 2016-11-11 (Actual)

PRIMARY OUTCOMES:
To assess recruitment rate to the study on first invitation | one year
To estimate proportion of recruited women who demonstrate willingness to wear the monitor two times | one year
  In light of investigator's previous work, no problems are anticipated in achieving 30 recruits in a year. However, study would be deemed successful if at least 80% of participants wear the monitor on second occasion and complete the study

SECONDARY OUTCOMES:
To measure success rate of fetal heart rate data across different stages of pregnancy | one year
  Success rate will be presented in percentage.

CONTACTS AND LOCATIONS:
Locations (1):
- Jessop Wing Hospital, Sheffield, United Kingdom

REFERENCES:
- [Background] Kapaya H, Broughton-Pipkin F, Hayes-Gill B, Loughna PV. Smoking in pregnancy affects the fetal heart: possible links to future cardiovascular disease. J Matern Fetal Neonatal Med. 2015;28(14):1664-8. doi: 10.3109/14767058.2014.964202. Epub 2014 Dec 15. PMID 25212975